CLINICAL TRIAL: NCT03939013
Title: Hepatitis C: Community Testing and Treatment (CT2 Study Myanmar)
Acronym: CT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: Myanmar Liver Foundation (Other); Foundation for Innovative New Diagnostics, Switzerland (Other); UNITAID (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT2/Alfred244-17/DMR2018-144
Record Dates: First submitted 2019-04-17; First posted 2019-05-06 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C
Keywords: hepatitis C; Myanmar; primary care; direct acting antivirals
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Access to point-of-care hepatitis C testing in community setting to facilitate hepatitis C treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xpert HCV VL, sof/dac (local standard of care therapy) (Experimental): Use of Cepheid GeneXpert HCV VL device as diagnostic tool to test for HCV RNA for diagnosis of chronic hepatitis C infection, for assessment of sustained virological response at 12 weeks post treatment completion
  Interventions: Diagnostic Test: Xpert HCV VL

INTERVENTIONS:
Diagnostic Test: Xpert HCV VL — Use of Cepheid GeneXpert HCV VL test as diagnostic tool to test for HCV RNA for diagnosis of hepatitis C infection, to test for sustained virological response at 12 weeks post treatment completion
  Other Names: Cepheid GeneXpert; Xpert HCV RNA

SUMMARY:
Implementation-effectiveness hybrid trial assessing acceptability, feasibility and cost-effectiveness of community-based point-of-care testing and treatment for hepatitis C. Utilises Cepheid GeneXpert HCV VL device as diagnostic tool (diagnosis of chronic infection and assessment of treatment outcome) and sofosbuvir/daclatasvir for HCV therapy (local standard of care).

DETAILED DESCRIPTION:
Historically, testing and treatment for hepatitis C has been confined to centralised laboratories and tertiary hospitals respectively. Recent advancements in point-of-care testing for hepatitis C (anti-HCV antibody and HCV RNA/VL) and treatment options with the introduction of direct acting antivirals allows for testing and treatment to occur in de-centralised primary care settings.

This study is an effectiveness-implementation hybrid study to assess the feasibility, acceptability, effectiveness and cost-effectiveness of a de-centralised approach to hepatitis C testing and treatment at community-based clinics in Yangon, Myanmar. Generalist doctors trained in hepatitis C treatment will prescribe direct acting antiviral therapy to eligible participants.

The study will utilise SD Bioline HCV RDT and Cepheid GeneXpert HCV VL test; and sofosbuvir/daclatasvir to treat hepatitis C. Test of cure will be performed at 12 weeks post-treatment completion to assess sustained virological response (SVR).

Study inclusion criteria prior to recruitment into study:

* Aged ≥18 years
* Attendance at study site
* Willing and able to provide written informed consent

Study exclusion criteria prior to recruitment into study:

* Confirmed HCV RNA positive result (chronic HCV infection) prior to study recruitment
* Treatment experienced (either DAA or pegylated interferon)
* Hepatitis B virus (HBV) infected
* Human Immunodeficiency Virus (HIV) infected
* estimated glomerular filtration rate (eGFR) <30
* Active tuberculosis (if known active tuberculosis or as per symptom screening assessment)
* Pregnant women
* Serious drug-drug interaction with sofosbuvir/daclatasvir of a drug that the patient is unwilling or unable to stop taking

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Attendance at study site
* Willing and able to provide written informed consent

Exclusion Criteria:

* Confirmed HCV RNA positive result (chronic HCV infection) prior to study recruitment
* Treatment experienced (either DAA or pegylated interferon)
* Hepatitis B virus (HBV) infected
* Human Immunodeficiency Virus (HIV) infected
* estimated glomerular filtration rate (eGFR) <30
* Active tuberculosis (if known active tuberculosis or as per symptom screening assessment)
* Pregnant women
* Serious drug-drug interaction with sofosbuvir/daclatasvir of a drug that the patient is unwilling or unable to stop taking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Proportion of Ab positive patients who receive GeneXpert HCV VL test | 6-9 months of recruitment
  Calculated by using Number of HCV Ab tests performed, Number of HCV RNA tests performed. Aggregate data is taken from patient-level case report forms recording results of tests performed (Clinical Case Report Form 1 & 2).
Proportion of RNA positive patients who receive direct-acting antiviral therapy for chronic hepatitis C infection | 9-12 months of recruitment & treatment
  Calculated by using Number of HCV RNA positive patients, Number of patients started on DAAs. Aggregate data is taken from patient-level case report forms recording results of tests performed and treatment plan (Clinical Case Report Form 1, 2 & 3).
Proportion of patients who complete direct-acting antiviral therapy for chronic hepatitis C infection | 9-18 months
  Calculated by using Number of patients started on DAAs, Number of patients who completed treatment. Aggregate data is taken from patient-level case report forms recording results of tests performed and treatment plan (Clinical Case Report Form 1, 2, 3, 4 & 5).
Proportion of patients who achieve SVR12 who started on direct-acting antiviral therapy for chronic hepatitis C infection | 9-18 months
  Calculated by using Number of patients started on DAAs, Number of patients who completed treatment, Number of patients who achieve SVR12 as measured by GeneXpert HCV VL not detected 12 weeks post completion of treatment. Aggregate data is taken from patient-level case report forms recording results of tests performed and treatment plan (Clinical Case Report Form 1, 2, 3, 4 & 5).

SECONDARY OUTCOMES:
Satisfaction of testing and treatment pathway among patients | 6-18 months
  Measured using a patient completed survey covering domains of satisfaction with care received, any barriers to accessing care and preferences for testing and treatment as per standard of care (hospital - prior experience) vs intervention (community based - trial experience).
Costing of testing and treatment pathway at community site | 6-18 months
  Measured using clinical workflow observations and costing tool; collecting data on staff time spent with patient on each phase of pathway, staff costs and consumables.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hellard, Principal Investigator — Burnet Institute; Hla Htay, Principal Investigator — Burnet Institute
Locations (2):
- Burma (2):
  - Myanmar Liver Foundation Than Sitt Charity Clinic, Yangon
  - Thingangyun Clinic, Yangon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Draper BL, Yee WL, Shilton S, Bowring A, Htay H, Nwe N, Markby J, Kyi KP, Easterbrook P, Naing W, Win TM, Aung KS, Howell J, Pedrana A, Hellard M. Feasibility of decentralised, task-shifted hepatitis C testing and treatment services in urban Myanmar: implications for scale-up. BMJ Open. 2022 May 3;12(5):e059639. doi: 10.1136/bmjopen-2021-059639. PMID 35504640